CLINICAL TRIAL: NCT00928031
Title: Collection of Long-Term Outcome Data for Subjects Who Have Previously Participated in Selected Ipilimumab (MDX-010) Studies in Metastatic Melanoma
Brief Title: Long-term Data Collection for Subjects in MDX-010 Studies
Acronym: MDX010-28
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Other Study IDs: MDX010-28
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to collect disease status and overall survival information for all Subjects in MDX-010 studies.

DETAILED DESCRIPTION:
This is a multicenter, follow-up study in up to 191 subjects with metastatic melanoma who were previously enrolled and treated in ipilimumab studies MDX010-02, MDX010-08, and MDX010-15. The purpose of this study is to 1) collect the date and cause of death, if known, for all deceased subjects who participated in any of the specified studies; 2) collect the date of progression for subjects who completed the studies with stable disease or better; and 3) prospectively follow all surviving subjects to determine progression-free and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who were previously enrolled in MDX-010 studies MDX010-02, MDX010-08, or MDX010-15.
2. Subjects (or if applicable, next of kin), who are alive at the time of contact must have read, understood, and provided written informed consent and health Insurance Portability and Accountability Act (HIPAA) authorization after the nature of the study has been fully explained.
3. For subjects who have died or have been lost to follow-up(the subject status at end of original ipilimumab study), approval from the appropriate site IRB, specifying or limiting appropriate means for obtaining information, must be granted prior to collection of any information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who received any dose of ipilimumab (MDX-010) in MDX010-02, MDX010-08, and MDX010-15 and were alive at the time of study completion.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2007-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Urba, MD PhD, Principal Investigator — Providence Health & Services
Locations (11):
- United States (11):
  - Arizona Cancer Center, Tuscon, Arizona
  - Pacific Shores Medical Group, Long Beach, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - USC Norris Cancer Center, Los Angeles, California
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - St. Francis Research Foundation, Beech Grove, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYU Cancer Institute, New York, New York
  - Carolinas Cancer Care, Charlotte, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - Huntsman Cancer Institute, Salt Lake City, Utah